CLINICAL TRIAL: NCT03335631
Title: A Preference-Based Trial of Two Exercise Delivery Methods in Men With PC on ADT
Brief Title: Preference-Based Exercise RCT for Men With PC on ADT
Acronym: PBExRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-5506
Record Dates: First submitted 2017-10-19; First posted 2017-11-08 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-supervised (Experimental): This intervention arm will include 3 group, supervised sessions per week for 6 months with a certified exercise specialist. Supervised sessions will be delivered in a group format with 4-8 participants per group. Flexibility training will include stretching for 5-10 minutes at the beginning and end of each session. Aerobic training will involve 30 minutes of low-impact step aerobics. Resistance training will be conducted using resistance bands, a stability ball, and an exercise mat with 8 prescribed exercises that target the major muscle groups. Participants will be encouraged to perform exercises independently on additional days, for a total of 4-5 days per week of exercise.
  Interventions: Behavioral: Exercise
- Home-based (Experimental): The same protocol and training frequency as the supervised programs described above will be followed. However, all exercises will be completed independently by participants. Specific exercises in the aerobic program may be modified to accommodate patient preference (same target heart rate range as the supervised group). Participants will be supported with smartphone technology and remote 'health coaches' during the intervention phase. This will help to ensure participant adherence, appropriate progression, and safety.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Moderate intensity mixed-modality exercise 4-5 days per week, with a target of 60 minutes per session.

SUMMARY:
Prostate cancer affects 1 in 7 men. Half of these men are treated with androgen deprivation therapy (ADT). ADT slows disease progression and prolongs survival, but it also leads to worse quality of life (QOL), fatigue, loss of strength and fitness, osteoporosis, and diabetes.

The investigators' recent research has shown that individually supervised exercise, supervised group exercise and home-based exercise are equally good at improving these side effects. Now the investigators are doing a larger trial with multiple centres to see whether supervised group or home-based exercise is clinically better and more economical.

A major challenge in such trials is that a significant number of men refuse to be randomized because (a) the participant lives too far from a study centre and cannot come for supervised exercise; or (b) the participant has a strong preference as to which type of exercise program the participant wants to do. Experts have raised concerns that classic randomized trials are too restrictive, selective, and less practical; the study results are less applicable to the real world. Despite its obvious importance, it is not known whether men who refuse to be randomized to an exercise trial but are otherwise willing to participate would benefit similarly to men who are randomized. In this study, we will recruit men who are otherwise eligible for our randomized trial but refuse it for one of the reasons above. We will allow these men to choose either supervised group or home-based exercise, and then compare them to the men who are being randomized to the two treatments in 3 important ways. First, are participants similar in terms of personal characteristics, QOL, and fitness levels? Second, do participants respond similarly to exercise in terms of QOL and physical fitness benefits? Third, do participants actually exercise as much as the randomized men? This work will help the research team understand whether there is a need to change the way exercise trials are done in order to be more relevant and wide-reaching for Canadians with a variety of health conditions.

DETAILED DESCRIPTION:
BACKGROUND: The backbone of scientific evidence to address most scientific questions, including behavioural interventions, is randomized controlled trials (RCTs). Prostate cancer is the most common malignancy in men, affecting 1 in 7 men. Almost 50% of these men will receive androgen deprivation therapy (ADT) at some point after diagnosis to reduce disease progression and prolong survival. ADT is associated with multiple adverse effects, including diminished quality of life (QOL), fatigue, reduced muscle mass, and metabolic effects. Numerous RCTs in the setting of men on ADT have demonstrated that exercise programs, particularly supervised 1:1 in-centre programs, are clinically effective. However, they are resource-intensive and have low scalability. Alternative delivery models such as group-based supervised exercise or home-based exercise are promising alternatives but require rigorous efficacy data. While conducting a two-centre exercise trial comparing different exercise delivery models, fewer than 40% of eligible men agreed to participate. Two common reasons why men declined participation were distance to exercise centres and unwillingness to be randomized. Novel clinical trial designs, such as preference-based trials, may help answer effectiveness questions and enhance generalizability by recruiting a more representative pool of men. Increased efficiencies in recruitment, however, may come at a cost of bias with non-randomized designs as well as differential effects of exercise and varying adherence. In parallel with a multi-centre phase III RCT funded by CIHR, we propose to conduct a pilot preference-based trial, examining 3 key issues. First, can we successfully enroll men who are unwilling to be randomized due either to distance from centre or a strong preference for one exercise delivery model? Second, are these men different from men who are randomized in terms of baseline characteristics, study retention, and adherence to the intervention? Third, are the benefits of an exercise program similar to men who are randomized to the same arm?

OBJECTIVES:

To determine, in men with PC on ADT who are otherwise eligible to participate in a RCT of different exercise delivery models but decline to be randomized due to distance from the study centre or strong preference for one exercise delivery model:

1. What proportion of these men is willing to be enrolled in a preference-based trial.
2. How comparable are baseline characteristics of men who agree to participate in the intervention arm of their choice and all those in the randomized study?
3. How comparable are study retention and adherence to the intervention for men in the corresponding arms of the preference based trial and randomized trial?
4. How comparable are the benefits in terms of quality of life (QOL) and physical fitness outcomes in those with a preference for a particular exercise and those without a preference?

HYPOTHESES

1. Systematic differences exist in baseline characteristics, specifically distance to the study centre, age, education, prior experience with participating in exercise programs, and fatigue severity among participants willing to be randomized versus not randomized to an exercise intervention.
2. Adherence will be greater among those selecting treatment by preference vs being randomized.
3. Benefits (QOL and fitness) will be greater among those selecting treatment versus being randomized.

METHODS: Patients aged 18 or older on ADT for high-risk/locally advanced, biochemically relapsed, or asymptomatic metastatic prostate cancer will be eligible if they are otherwise eligible for an ongoing phase III RCT of exercise but decline to participate due to either distance from study centre or strong preference for one exercise delivery model. The main phase III RCT is examining a 6-month individualized, progressive, mixed-modality exercise program including aerobic, resistance, and flexibility components delivered using one of two delivery models: supervised in-centre group exercise 3 times weekly or home-based exercise supported by a Fitbit, smart phone app, and remote health coach.

To meet the objectives of this pilot preference trial, we will enroll 50 men per preference arm at three experienced study sites (Princess Margaret Cancer Centre, Toronto, Scarborough and Rouge Hospital, Scarborough and the University of Calgary, Calgary and). Aim 1. We will report the proportion of men who are eligible for the preference-based trial who agree to participate, overall and by treatment arm and reason for refusal to be randomized.

Aim 2/Hypotheses 1 and 2. We will compare the participants in the preference-based trial to those in the RCT. Comparisons of baseline characteristics will be between the total number of participants in the RCT compared separately to each arm of the preference trial. ANOVA will be used for continuous variables and chi-square analysis for categorical variables. Variables to be compared include distance from participants' home to the study centre, age, education, prior participation in an exercise program, and symptom severity. Differences will be presented with 95% CIs.

Aim 3/Hypothesis 3. Within-group change scores will be assessed for the preference-based groups, and the mean changes along with the 95%CIs will be reported. Next, we will compare these changes for the co-primary and secondary outcomes between the preference-based groups and the phase III RCT (e.g., combined preference arms to combined RCT arm) to obtain the so-called selection-effect. Finally, although it is subject to confounding by unknown preference effects in the RCT participants, we will estimate the differences between outcomes in those randomized to and choosing each specific exercise delivery method, using constrained linear mixed effects model adjusting for the baseline value and ADT duration. Skewed data will be transformed as appropriate.

SIGNIFICANCE: Behavioural interventions require significant patient commitment and although most RCTs to date have shown evidence of benefit on various outcomes, recruitment rates have been low and many otherwise eligible men are not willing to be randomized for different reasons. Designing trials that allow inclusion of such men is obviously going to improve generalizability but whether the results of interventions are similarly effective and understanding the feasibility and potential biases of enrolling such men are fundamental unresolved issues. This pilot study will take advantage of an existing trial to begin to answer these questions and determine whether a larger preference-based trial is worth undertaking. Our findings have potential widespread implications for behavioural trials across many health care settings.

ELIGIBILITY:
Inclusion Criteria:

* men with histologically confirmed PC who are starting or continuing on ADT for at least 6 months
* fluent in English,
* able to provide consent.

Exclusion Criteria:

* already meeting guidelines for moderate to vigorous physical activity (MVPA)
* conditions that would interfere with ability to participate

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy-Fatigue (FACT-F) scale over time | Baseline, 3, 6, 12 months
  The FACT-F is a questionnaire that includes 13 items measuring cancer-related fatigue.
  Total Score Range = 0-52 (higher score = lower fatigue)
Change in 6 minute walk test (6MWT) scores over time | Baseline, 3, 6, 12 months
  The 6MWT is a commonly used, validated measure that assesses functional endurance.

SECONDARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy-General (FACT-G) scale over time | Baseline, 3, 6, 12 months
  The FACT-G is a questionnaire that is well-validated and widely used to measure quality of life (QOL).
  Total Score Range = 0-108 (higher score = higher QOL)
Change in Functional Assessment of Cancer Therapy-Prostate (FACT-P) scale over time | Baseline, 3, 6, 12 months
  The FACT-P is a questionnaire that supplements the FACT-G with 12 prostate-specific items covering domains of urinary function, sexual function, pain, and related symptoms.
  Range = 0-48 (higher score = fewer prostate-specific symptoms)
Change in 5 Timed Chair Stand Test over time | Baseline, 3, 6, 12 months
  A common, simple, and validated measure of functional lower body strength.
Change in grip strength using a Jamar dynamometer over time | Baseline, 3, 6, 12 months
  Grip strength is a measure of upper body strength and predicts long-term disability and mortality in middle-aged and older adults.
Change in body composition (fat mass, fat free mass, and body fat percentage) measured via body impedance analysis (BIA) over time | Baseline, 6, 12 months
  Body composition will be measured using bioelectrical impedance analysis (BIA).
Change in fasting lipids over time | Baseline, 6, 12 months
  Fasting lipids will be measured.
Change in blood glucose over time | Baseline, 6, 12 months
  Blood glucose will be measured.
Change in glycated hemoglobin over time | Baseline, 6, 12 months
  Glycated hemoglobin will be measured.
Change in hemoglobin over time | Baseline, 6, 12 months
  Hemoglobin will be measured.
Change in prostate specific antigen (PSA) over time | Baseline, 6, 12 months
  Prostate-specific antigen (PSA) will be measured.
Change in weekly minutes of moderate-vigorous physical activity (MVPA) over time | Baseline, 3, 6, 12 months
  Accelerometry will be used to measure weekly minutes of MVPA as an indicator of adherence at each time point.
Change in Health Care Climate Questionnaire (HCCQ) over time | Baseline only
  The Health Care Climate Questionnaire (HCCQ short form) assess participant perceptions of their health care team.
  Range = 0-7 (higher = better)
Change in Behavioral Regulations in Exercise Questionnaire-2 (BREQ-2) over time | Baseline, 6, 12 months
  Behavioral Regulations in Exercise Questionnaire-2 (BREQ-2) is a validated questionnaire that assess predictors of adherence.
  Comprised of 4 subscales:
  External regulation, range = 0-4 (higher = better) Introjected regulation, range = 0-4 (higher = better) Identified regulation, range = 0-4 (higher = better) Intrinsic regulation, range = 0-4 (higher = better)
Change in Psychological Need Support and Frustration Scale - Relatedness Items (PNSF - Relatedness Items) over time | Baseline, 6, 12 months
  The Psychological Need Support and Frustration Scale - Relatedness Items will be used to measure relatedness.
  Total Score Range = 1-5 (higher = better)
Change in Planning, Attitudes, & Barriers scale over time | Baseline, 6, 12 months
  The Planning, Attitudes, & Barriers (PAB) scale is a validated questionnaire that will be used to assess the likelihood of exercise behavior and adherence over time.
  Comprised of 11 subscales:
  Attitudes subscale, range = 1-7 (higher = better); Support subscale, range = 1-7 (higher = better); Motivation subscale, range = 1-7 (higher = better); Intentions subscale, range = 1-7 (higher = better); Planning subscale, range = 1-7 (higher = better); Disease/treatment influences subscale, range = 1-7 (higher = better); Disease/treatment frequency subscale, range = 1-7 (higher = better); Life-related influences subscale, range = 1-7 (higher = better); Life-related frequency subscale, range = 1-7 (higher = better); Motivated-related influences subscale, range = 1-7 (higher = better); Motivated-related frequency subscale, range = 1-7 (higher = better) Note: No total score is derived from this questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir MH Alibhai, MD, MSc, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - University of Calgary/Tom Baker Cancer Centre, Calgary, Alberta
  - Scarborough and Rouge Hospital, Scarborough Village, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alibhai SMH, Papadopoulos E, Durbano S, Tomlinson G, Mina DS, Ritvo P, Sabiston CM, Matthew AG, Chiarotto J, Sidani S, Culos-Reed SN. Preference-based versus randomized controlled trial in prostate cancer survivors: Comparison of recruitment, adherence, attrition, and clinical outcomes. Front Oncol. 2022 Dec 12;12:1033229. doi: 10.3389/fonc.2022.1033229. eCollection 2022. PMID 36578945